CLINICAL TRIAL: NCT05371028
Title: A Non-interventional, Multicentre Retrospective Study of the Effectiveness and Safety of Teduglutide (REVESTIVE®) in Short Bowel Syndrome Patients in Canada
Brief Title: A Study of Teduglutide (Revestive®) in Participants With Short Bowel Syndrome (SBS) in Canada
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-4006; MACS-2020-112501 (Other: Takeda)
Record Dates: First submitted 2022-04-28; First posted 2022-05-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Short Bowel Syndrome (SBS)
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With SBS-IF: Participants with SBS-IF who as part of standard or routine clinical practice, must have received teduglutide (Revestive®) treatment and were dependent on parenteral support prior to teduglutide treatment initiation will be observed in this retrospective observational study for up to 48 months.
  Interventions: Other: Non-interventional Study

INTERVENTIONS:
Other: Non-interventional Study — This is non-interventional study.

SUMMARY:
The main aim of this study is to assess the effectiveness and side effects of teduglutide (Revestive®) in real-world clinical practice setting in adult participants with intestinal failure due to short bowel syndrome (SBS-IF) in Canada.

This study is about collecting existing data only; participants receive teduglutide (Revestive®) by their doctors according to the clinical practice but not as part of this study. No new information will be collected during this study.

The study will be conducted using data from the Takeda OnePath Patient Support Program (PSP) or Takeda Global Pharmacovigilance.

ELIGIBILITY:
Inclusion criteria:

* Participants more than or equal to (>=) 18 years of age at first dose of teduglutide diagnosed with intestinal failure due to short bowel syndrome as a result of intestinal resection. Note: As "SBS as result of major intestinal resection" is a criterion for teduglutide treatment reimbursement, it is assumed that all participants receiving teduglutide in the PSP have SBS-IF as a result of intestinal resection.
* Stable participants with SBS-IF who were dependent on parenteral support prior to teduglutide treatment initiation, and were treated with teduglutide during the study period with at least 6 months of follow-up data available before the end of the study period.
* Participants who have provided informed consent for secondary use of data for research.

Exclusion criteria:

- Participants with active gastrointestinal malignancy OR a history of gastrointestinal malignancy in the past 5 years before start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with SBS-IF, who were treated with teduglutide (Revestive®) in Canada will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Weekly Volume of Parenteral Nutrition (PN)/Intravenous (IV) Fluid Requirement at Week 24 | Baseline and at Week 24
  Weekly volume of PN/IV fluid requirement at baseline before teduglutide treatment and at Week 24 after initiation of teduglutide treatment will be reported.
Average Change in Number of Days per Week With PN/IV Usage | 6 months before teduglutide treatment initiation and 6 months after teduglutide treatment initiation (approximately 12 months
  Average change in number of days per week with PN/IV usage in the 6 months before teduglutide treatment initiation and 6 months after teduglutide treatment initiation will be reported.
Percentage of Participants Achieving PN/IV Independence During the Study Period | Up to 48 Months
  Percentage of participants who will achieve PN/IV independence during the study period will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Weekly Volume of PN/IV Fluid Requirement | Baseline and at 6, 12, 24, 36 and 48 months after initiation of teduglutide treatment
  Change from baseline in weekly volume of PN/IV fluid requirement at 6,12, 24, 36 and 48 months after initiation of treatment with teduglutide will be reported.
Number of Participants Achieving Response of 20 percent (%) to 100% Reduction From Baseline in Weekly Parenteral Support (PS) Volume | Up to 48 months after teduglutide treatment initiation
  Number of participants achieving response of 20% to 100% reduction from baseline in weekly PS volume will be reported.
Percentage of Participants Achieving 20 % to 100% Reduction From Baseline in Weekly Parenteral Support (PS) Volume | Baseline and at 6, 12, 24, 36 and 48 months after initiation of teduglutide treatment
  Percentage of participants achieving 20% to 100% reduction from baseline in weekly PS volume at 6, 12, 24, 36 and 48 months after initiation of treatment with teduglutide will be reported.
Change From Baseline in Number of Days per Week With PN/IV Usage | Baseline and at 6, 12, 24, 36 and 48 months after initiation of teduglutide treatment
  Change from baseline in number of days per week with PN/IV usage at 6,12, 24, 36 and 48 months after teduglutide treatment initiation will be reported.
Number of Participants With Reasons of Treatment Interruption and Discontinuation | From teduglutide treatment initiation up to 48 months
  Number of participants with reasons of treatment interruption and discontinuation will be reported.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From treatment initiation up to 6 months after teduglutide treatment discontinuation (approximately 48 months)
  An AE is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. A SAE is any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Innomar Strategies, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/7a0519256a734775?idFilter=%5B%22TAK-633-4006%22%5D